CLINICAL TRIAL: NCT06239610
Title: DrIFT 2 Study: Displacement in Feeding Tubes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parkview Health (Other)
Responsible Party: Principal Investigator, Danielle Payne, FNP, Clinical Nurse Researcher & Nursing Research Program Coordinator, Parkview Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NUR23-1127DrIFT2
Record Dates: First submitted 2024-01-05; First posted 2024-02-02 (Actual); Results first posted 2025-07-24 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Enteral Nutrition
Keywords: feeding tube; coretrak; tube migration; critical care; enteral nutrition; gastric tube feeding

STUDY DESIGN:
Intervention Model Description: longitudinal, repeated measures design replication study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- feeding tube migration (Other): Use of an EMPD to assess for FT migration in all eligible critical care patients requiring the use of a feeding tube during admission.
  Interventions: Device: electromagnetic placement device

INTERVENTIONS:
Device: electromagnetic placement device — Daily use of an EMPD to verify FT position
  Other Names: Cortrak* 2 Enteral Access System

SUMMARY:
The proposed study will use an electromagnetic placement device (EMPD), Cortrak* 2 Enteral Access System (EAS™), Avanos Medical, to verify feeding tube (FT) position on a daily basis to assess for migration. The EMPD provides real-time FT placement data. A sensor located on the distal end of the FT guidewire communicates with a receiver unit which sits on the patient's abdomen. Three visual insertion tracings with varying views (anterior, lateral, and depth/cross-section) can be saved and printed for comparison.

DETAILED DESCRIPTION:
Two previous studies have been completed with similar methodology. A pilot study of 50 subjects was performed using the original Cortrak* (2 insertion views) and found only minimal forward migration. No reverse migration was reported in one study.

A pilot study of 20 patients with 62 feeding tube assessment identified 8 migration events (5 retrograde and 3 forward), these events only occurred within the small bowel. Based on this data, a recommendation could be made that there is no need to check feeding tube placement routinely every four hours. However, due to the small sample size, additional research is needed to confirm this finding. It is also unknown if there may be more migration with positioning changes, for example, up in the chair or prone position.

The proposed study will use an electromagnetic placement device (EMPD), Cortrak* 2 Enteral Access System (EAS™), Avanos Medical, to verify FT position on a daily basis to assess for migration. The proposed study will take place in critical care units at Parkview Health. The primary aim will be to determine if replication of the pilot study results in similar findings. Investigators will also explore other factors that may be associated with FT migration, such as patient mobility (ambulation or sitting at bedside or prone position) and transporting out of the critical care unit for diagnostic procedures. Researchers anticipate that results from this study will provide a better understanding of FT position and migration over time and ultimately influence recommendations for practice for frequency of routine FT verification. Standard of care for assessing feeding tube placement location every 4 hours will remain in place. The study will add an additional assessment for feeding tube location daily. This study will expand on the findings from the initial pilot study with a larger sample size.

ELIGIBILITY:
Inclusion Criteria:

* Adult critical care patients with small bore feeding tube inserted within last 24-48 hours
* Initial Cortrak insertion tracings: all 3 views available
* Cortrak guidewire available

Exclusion Criteria:

* Unable to speak or understand English language
* Pregnancy
* Prisoners
* FT anticipated to be removed within 24 hours
* Contraindications to placing a mark on the abdomen for top foot of receiver unit (large dressings, open abdomen, halo vest, etc.)
* Original guidewire unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-08-11 (Actual); Study Completion 2024-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan R Powers, Principal Investigator — Parkview Health
Locations (1):
- Parkview Regional Medical Center, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
A data sharing agreement is in place stipulating that data provided to Data Recipient will not contain any "Protected Health Information" (as that term is defined in the HIPAA privacy rule at 45 C.F.R. §160.103) and shall be de-identified in accordance with 45 C.F.R. §164.514(b) of the HIPAA privacy rule. he Parties agree that the Data will be completely De-Identified.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will become available after data cleaning and analysis, which is anticpated to be 10 months.
Access Criteria: All data will be de-identified and in aggregate format.

REFERENCES:
- [Background] Metheny NA, Stewart BJ, McClave SA. Relationship between feeding tube site and respiratory outcomes. JPEN J Parenter Enteral Nutr. 2011 May;35(3):346-55. doi: 10.1177/0148607110377096. PMID 21527596
- [Background] Initial and Ongoing Verification of Feeding Tube Placement in Adults (applies to blind insertions and placements with an electromagnetic device). Crit Care Nurse. 2016 Apr;36(2):e8-e13. doi: 10.4037/ccn2016141. No abstract available. PMID 27037348
- [Background] Bourgault AM, Heath J, Hooper V, Sole ML, Nesmith EG. Methods used by critical care nurses to verify feeding tube placement in clinical practice. Crit Care Nurse. 2015 Feb;35(1):e1-7. doi: 10.4037/ccn2015984. PMID 25639583
- [Background] Metheny NA, Stewart BJ, Mills AC. Blind insertion of feeding tubes in intensive care units: a national survey. Am J Crit Care. 2012 Sep;21(5):352-60. doi: 10.4037/ajcc2012549. PMID 22941709
- [Background] Milsom SA, Sweeting JA, Sheahan H, Haemmerle E, Windsor JA. Naso-enteric Tube Placement: A Review of Methods to Confirm Tip Location, Global Applicability and Requirements. World J Surg. 2015 Sep;39(9):2243-52. doi: 10.1007/s00268-015-3077-6. PMID 25900711
- [Background] Kearns PJ, Donna C. A controlled comparison of traditional feeding tube verification methods to a bedside, electromagnetic technique. JPEN J Parenter Enteral Nutr. 2001 Jul-Aug;25(4):210-5. doi: 10.1177/0148607101025004210. PMID 11434652
- [Background] Metheny N, McSweeney M, Wehrle MA, Wiersema L. Effectiveness of the auscultatory method in predicting feeding tube location. Nurs Res. 1990 Sep-Oct;39(5):262-7. PMID 2119031
- [Background] Makic MB, Martin SA, Burns S, Philbrick D, Rauen C. Putting evidence into nursing practice: four traditional practices not supported by the evidence. Crit Care Nurse. 2013 Apr;33(2):28-42. doi: 10.4037/ccn2013787. PMID 23547123
- [Background] Bourgault AM, Powers J, Aguirre L, Hines R. Migration of Feeding Tubes Assessed by Using an Electromagnetic Device: A Cohort Study. Am J Crit Care. 2020 Nov 1;29(6):439-447. doi: 10.4037/ajcc2020744. PMID 33130862
- [Background] Bourgault AM, Aguirre L, Ibrahim J. Cortrak-Assisted Feeding Tube Insertion: A Comprehensive Review of Adverse Events in the MAUDE Database. Am J Crit Care. 2017 Mar;26(2):149-156. doi: 10.4037/ajcc2017369. PMID 28249868
- [Background] Bourgault AM, Deb C, Aguirre L, Xie R, Rathbun KP, Sole ML. Microbiome profile informs cleansing and storage practices for reusable feeding tube stylets in critical care. Nutr Clin Pract. 2023 Apr;38(2):411-424. doi: 10.1002/ncp.10904. Epub 2022 Aug 19. PMID 35985807
- [Background] Wang MC, Chang SH. Nonparametric Estimation of a Recurrent Survival Function. J Am Stat Assoc. 1999 Mar 1;94(445):146-153. doi: 10.1080/01621459.1999.10473831. PMID 24244058

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient was removed due to a missing feeding tube stylet.
Period: Overall Study
Arm/Group | Feeding Tube Migration
Started | 119
Completed | 108
Not Completed | 11
Not completed — no usable migration data for minimum of one day | 11

BASELINE CHARACTERISTICS:
Arm/Group | Feeding Tube Migration
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 50
  >=65 years | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The 12 patients, who could not be included due to only having one day of FT zone data, were reviewed for reasons of withdrawal. Five (42%) of these patients had unexpected withdrawal of care due to family decisions or hospice admission. Four patients had their FTs removed during ETT extubation. Two patients improved significantly and were able to start an oral diet. One patient was removed due to a missing feeding tube stylet.
  years | 63.92 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 61
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 108
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.96 (8.42)

OUTCOME MEASURES:

1. Primary Outcome: Tube Migration
Description: Number of participants with clincially significant feeding tube retrograde migration
Time Frame: 5 days or until FT removed, whichever came first
Measure: Count of Participants; unit: Participants
Arm/Group | Feeding Tube Migration
Number analyzed (Participants) | 108
Participants | 6

2. Primary Outcome: Effect of ETT Extubation on FT Movement
Description: Number of participants with clincially significant retrograde migration after extubation
Time Frame: 5 days or until FT removed, whichever came first
Population: Total number of participants in study (n=108) who were intubated 30/108.
Measure: Count of Participants; unit: Participants
Arm/Group | Feeding Tube Migration
Number analyzed (Participants) | 30
Participants | 2

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Feeding Tube Migration
All-Cause Mortality (participants affected / at risk) | 0/119
Serious Adverse Events (participants affected / at risk) | 0/119
Other Adverse Events (participants affected / at risk) | 0/119

LIMITATIONS AND CAVEATS:
This study occurred at a single study site with a small sample size. Multisite and larger sample size studies would increase the confidence around the size of our estimated effects and may also identify different factors associated with migration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT06239610/Prot_SAP_000.pdf